CLINICAL TRIAL: NCT03009513
Title: Teneligliptin-Glimepiride DDI Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP_C103
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: Teneligliptin+Glimepiride

INTERVENTIONS:
Drug: Teneligliptin+Glimepiride

SUMMARY:
An open label, one sequence study to investigate the pharmacokinetic drug interaction between Teneligliptin and Glimepiride in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adult aged 20 to 45 years
2. Body weight ≥ 50kg, and BMI between 18 and 29 kg/m2 at screening
3. Subject who agrees to use a medically acceptable double-barrier method of contraception and not to donate sperms from the first dose until 2 months after the last dose.
4. Subject who was given, and fully understood, the information about the study, and has provided voluntary written informed consent to participate in the study and agreed to comply with the study requirements.

Exclusion Criteria:

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 24hr
Area under the plasma concentration versus time curve (AUC) | 24hr